CLINICAL TRIAL: NCT04670250
Title: The Validity of Novel Non-invasive Inflammatory Markers for Monitoring of Patients With Ulcerative Colitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed Kamal Eldin Mohammed Ali, assistant lecturer, Assiut University
Other Study IDs: non invasive markers in IBD
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: IBD, Non Invasive Markers,IL6,Lactoferrin,Ferritin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newly diagnosed patients with ulcerative colitis: patients who are newly diagnosed to have ulcerative colitis who are above 18 years old,not pregnant and not known to have cancer colon
  Interventions: Diagnostic Test: non invasive markers

INTERVENTIONS:
Diagnostic Test: non invasive markers — non invasive markers (IL6, serum ferritin, fecal lactoferrin) used for monitoring of newly diagnosed patients with ulcerative colitis

SUMMARY:
Ulcerative Colitis (UC) is a disease known for repeated relapses and remissions. So, meticulous follow-up is required to individualize treatment plans according to the status of each patient. The currently used investigations are invasive, costy, and carry the risk of several side effects, making it difficult for the patient to adhere to his continuous follow-up.

Aim: To evaluate the viability of fecal lactoferrin, serum ferritin, and IL6 as noninvasive markers for detecting the activity and follow-up the patients of ulcerative colitis during remission.

DETAILED DESCRIPTION:
Introduction: Ulcerative Colitis (UC) is a disease known for repeated relapses and remissions. So, meticulous follow-up is required to individualize treatment plans according to the status of each patient. The currently used investigations are invasive, costy, and carry the risk of several side effects, making it difficult for the patient to adhere to his continuous follow-up.

Aim: To evaluate the viability of fecal lactoferrin, serum ferritin, and IL6 as noninvasive markers for detecting the activity and follow-up the patients of ulcerative colitis during remission.

Patients and Methods:

This is a prospective cohort study will include 160 patients. The study will be aMulticenterthat will be held in different Egyptian governorates. The patient must be, firstly, confirmed to be an ulcerative colitis patient by complete physical examination, laboratory evaluation by fecal calprotectin and CRP. Also, colonoscopy will be done for all included patients and they will be classified according to the Modified Mayo Endoscopic Score (MMES). Biopsies will be taken to confirm the diagnosis with histopathological examination. Fecal lactoferrin, S ferritin, and IL6 (the investigated markers) will be conducted for patients with confirmed diagnosis with UC. . All investigations, including colonoscopy, will be done once again after 3 months to follow up the included patients. The results of all tests will be correlated to the clinical and endoscopic findings of included patients to detect a cut off values to be used during remission and activity.

ELIGIBILITY:
Inclusion Criteria:

- Patients who are newly diagnosed to be ulcerative colitis. Patients >18 years old.

Exclusion Criteria:

* Patients who are >18 years old. Pregnant patients . Patients with colonic malignancies.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All newly diagnosed patients with ulcerative colitis will be included in the study
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The Validity of Novel Noninvasive Inflammatory Markers for Monitoring of Patients with Ulcerative Colitis. | 18 months
  the outcome will be to replace an invasive method used frequently to evaluate patients with ulcerative colitis like colonoscoy with a non invasive safe and hopfelly accurate method like fecal